CLINICAL TRIAL: NCT00548379
Title: The Effect of Vitamin D Supplementation on the Incidence of Pneumonia in Children in Afghanistan: a Randomized Controlled Trial
Brief Title: Kabul Vitamin D Supplementation Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); Aga Khan Health Services (Other); Aga Khan University (Other); Maywand Hospital, Kabul (Unknown)
Responsible Party: Semira Manaseki-Holland BMSci MBBS MFPHM MRCP MSc PhD, Chief Executive Officer for Central Asia,, Aga Khan Health Services, Afghanistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1963; WT082476MA
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Pneumonia; Vitamin D Deficiency
Keywords: vitamin D; pneumonia
MeSH Terms: conditions — Pneumonia; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Vitamin D
  Interventions: Drug: vitamin D
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vitamin D — vitamin D 100,000 units once in 3 months
  Arms: 1
Drug: placebo — olive oil 1ml
  Arms: 2

SUMMARY:
Background: Pneumonia is the leading cause of childhood mortality, accounting for 19% of the 10.6 million deaths that occur each year1. Case-control studies from Ethiopia2 and India3 suggest that sub-clinical vitamin D deficiency may increase ten times the risk of pneumonia in children. We postulate that controlling childhood vitamin D deficiency has the potential to dramatically reduce the incidence of pneumonia and save >700,000 lives each year since vitamin D deficiency is widespread in developing countries.

Aim: To investigate whether 3-monthly oral supplementation of 100,000iu vitamin D reduces pneumonia and its consequences among children aged 1-12 months (followed for 18 months), living in a deprived area of Kabul, Afghanistan, where >70% of young children are vitamin D deficient (<8ng/dl). The effect of vitamin D on the incidence of other diseases, in particular diarrhea and rickets will also be investigated.

Methods: Randomised double-blind placebo-controlled trial: 3000 children will be randomised to receive either 6 doses of vitamin D or placebo. The first dose will be given at the start of autumn and the second and subsequent doses every 3 months thereafter; children will be followed for 18 months. Incidence of pneumonia will be ascertained though weekly home visits (active surveillance) and from attendances and admissions at the trial clinic and wards in the hospital serving the study area (passive surveillance).

DETAILED DESCRIPTION:
Vitamin D, an essential micronutrient has a biological function in the formation and maintenance of strong bones. Vitamin D may help maintain a healthy immune system. In vitro studies have shown that 1,25-dihydroxyvitamine D3 (1,25(OH)2D3), the active metabolite of vitamin D is important for promoting and regulating immune responses. 1,25(OH)2D3 is an immune system modulator and induces expression of the TLR co-receptor CD145. 1,25(OH)2D3 directly induces antimicrobial gene expression an activity points to important therapeutic uses in treatment of opportunistic and some antibiotic resistant infections. Sub-clinical vitamin D deficiency has been associated with an increased risk of tuberculosis in adults through modification of polymorphisms in the vitamin D receptor. Vitamin is acquired primarily from sunlight; ultraviolet rays trigger synthesis in the skin, which is reduced in darker skins. The required UV light also reduces with distance from the equator to zero at latitudes above 500 in winter. Vitamin D deficiency can cause rickets, a common problem in many developing countries; prevalences of 5 to 45% in under-5 year old children have been found, even in places with abundant sunlight. Pneumonia is the leading cause of childhood mortality, accounting for 19% of the 10.6 million deaths that occur each year. Hospital-based case-control studies from Ethiopia and India suggest that vitamin D deficiency may substantially increase the risk of severe pneumonia in young children. High rates of vitamin D deficiency have also been found among children admitted to hospital for pneumonia, ranging from 43% in Tehran and Kuwait 27 to 50% in Yemen. Afghanistan has a very high under-5 and infant mortality (257 and 165 deaths/1000 live births respectively), and pneumonia is a leading cause of death in children. Women and young children have little exposure to sunlight, and thus are at risk of vitamin D deficiency. Women do not travel out of the home regularly; wear burkas or clothing that covers all but their hands and face. Swaddling of infants reduces exposure to sunlight, as does keeping young children in the mother's vicinity indoors. A survey during the winter of 2005 confirmed very high levels of vitamin D deficiency among young children in Kabul.

Controlling this deficiency has the potential to dramatically reduce the incidence of pneumonia and by so doing save lives. Three-monthly oral doses of 100,000iu of vitamin D have been proven to be safe and effective in alleviating vitamin D deficiency in high risk normal or rackettic children. Thus we propose to conduct a randomized controlled trial (RCT) in Afghanistan to test this.

Study area:

The trial will be carried out in District 1,2,3,7 and 8 of Kabul (latitude 34.280 N), where the vitamin D deficiency prevalence study was conducted in 2005. Most of these are old parts of Kabul with narrow, shaded lanes often with roofed tops between high walled mud houses; most houses have small courtyards with high walls so that for much of the day sunshine does not reach the courtyard. The population is socio-economically deprived with large families (5-10 children).

Recruitment:

Community sensitisation will be conducted through community and religious leaders and through public meetings. Recruitment will proceed in all streets of the chosen area which is within the catchment area of the study and continue house to house along each of those streets until 3000 children are recruited; 40 female Fieldworkers in pairs will recruit an average of 6 to 10 children per day over a 1-month period.

Informed consent:

At recruitment the Fieldworker will explain to the family the purpose of the study, the benefits offered and the procedures involved. An information sheet with the details of the study objectives, procedures, risk and benefits will also be given to the parents. Informed consent will then be obtained from both the mother and father of the child: finger prints and signature (literacy rate estimated at <50%) will be obtained in the presence of two witnesses, one a friend or family member and one the second Fieldworker.

Baseline data:

At recruitment and at regular periods throughout the study, Fieldworkers will collect data on a range of socio-economic and demographic variables, as well as the known risk factors for pneumonia or vitamin D deficiency, including exposure to cigarette smoke, type of fuel, vaccination, supplementation, diet/breastfeeding, and sun exposure.

Dosing/intervention and period:

6 doses of 100,000iu of vitamin D, or placebo, will be given by Fieldworkers during the first weekly home visit following recruitment and 3, 6, 9, 12 and 15 months later. If a child has vomiting at the time of supplementation, the Fieldworker will return weekly and dose after symptoms have subsided.

Randomization and packaging of intervention/placebo:

An independent statistician will produce the randomization list allocating individual study numbers to vitamin D or placebo within variable blocks of study numbers. This list will be used by the sourcing Pharmacy Department of AKU Hospital in Karachi to produce individual single dose sealed 1ml syringes for each child labeled with one study number. There will be no characteristics that would distinguish vitamin D dissolved in olive oil from the olive oil placebo in the syringes; there are no known side-effects that will distinguish those taking vitamin D from placebo.Oil from the syringes will be dropped in the mouth of each child at dozing. During the dosing weeks, Fieldworkers will receive 10 syringes each day with consecutive study numbers to be used that day and checks will be conducted in the evening. Thus Fieldworkers will only ever have 10 single doses in their possession, minimizing the possibility of mis-dosing.

Home visits (active case finding follow-up):

For 18 months and every 2 weeks, Fieldworkers will collect information on signs and symptoms of acute respiratory infections and diarrhea in the last 14 days, current breastfeeding status and vital status of study children. They will also be trained to take the child's temperature, count the respiratory rate twice using a UNICEF respiratory rate stop watch, examine for lower chest wall indrawing, look for dehydration and refer to the study clinic as appropriate. The causes of death occurring at home will be ascertained using a verbal autopsy.

Outpatient clinic and hospital admissions of pneumonias:

The first port of call will be a trial outpatient clinic set up within the Maywand Teaching Hospital located in the study area and within easy reach for all recruited families. This will be run by 4 paediatricians, who will receive refresher training in the diagnosis of pneumonia; they will work a shift system covering 24 hours, 7 days a week. They will be supervised by 1 senior paediatrician and he/she also will examine randomly a sample of other children seen at the clinic. The paediatricians will fill out a detailed clinical assessment form for each child, conduct pulse oximetry, request X-rays and treat (according to standard IMCI) 35 and/or refer for admission if there is severe pneumonia. The trial will cover costs of all IMCI recommended or hospital inpatient related ALRI medications.

Outcomes:

The primary outcome of the study is radiologically confirmed first or the only episode of pneumonia according to the WHO standard classification, i.e. [presence of dense or fluffy opacity that occupies a portion or whole of a lobe or the entire lung] or [presence of fluid in the lateral pleural space, between the lung and chest wall or both] 36. X-rays will be read by independent expert radiologists, blind to the child's allocation and clinical condition, and using a WHO Proforma Standardised Interpretation 36,37 of chest radiographs for the diagnosis of pneumonia in children.

The secondary outcome will be:

(1) Moderate or severe ALRI (using IMCI criteria) (2) Moderate or severe diarrhea (history of loose stools >3 times per day and history of oral rehydration or intravenous fluid therapy) (3) Incidence of hospital admissions for any illness; (4) Anthropometric indices at 0, 6, 12, 18 months (weight for height, weight for age, and height for age, head circumference) (5) All cause mortality and pneumonia specific mortality; (6) Biochemical markers of vitamin D deficiency [proportion of children with 25-OHD3 (cholicalciferol) <8ng/ml]38 at week 6 post vitamin D doses three (mid-spring) and four (mid-summer) in a random sample of 50 children each from the intervention and placebo group [We assume that the proportion of children with vitamin D deficiency will be 60% in the placebo group and it will be reduced to 30% in the intervention group at post vitamin D doses 3 and 4.]; (7) Pharmacodynamics of vitamin D supplementation will be determined by measuring serum 25-OHD3 (cholicalciferol) at day 2, week 6 and week 12 post vitamin D dose one in a random sample of 50 children each from the intervention and placebo groups] (8) The Thacher Radiological Score of Rickets 1 through wrist radiography of 10% random sample of children at the end of the 18 month follow up period.

Additional informed consent will be obtained for collecting blood samples. The sub-samples of children for measuring vitamin D level will be selected by the independent statistician. Venous blood samples will be taken at home by an experienced paediatric phlebotomist, and transported to the trial laboratory at the end of each morning and afternoon in clotted sampling bottles inside vaccine cool-boxes containing ice-packs. They will be centrifuged by experienced and retrained technicians and the extracted plasma frozen and stored at <20◦◦C At the end of the trial all frozen samples will be transported to the AKU Micronutrient Research Laboratory in Karachi for high 4 pressure liquid chromatography (HPLC) to establish vitamin D status.

Sample size:

We estimate that the incidence of acute lower respiratory infections (ALRI) in the placebo group will be 0.065/child /year 39 and 12% of the ALRI will be pneumonia 1. We assume that 25% of pneumonias will be repeat episodes during the 18 month follow up period. Thus the incidence of the first or the only episode of pneumonia in the placebo group will be 0.0585/child/year (0.65*0.12*0.75). We expect a 35% reduction in the incidence of pneumonia in the vitamin D group given that 73% of children have vitamin D deficiency in the study area and that the incidence of pneumonia is 10 times higher in vitamin D deficient children than in normal children 18, 26. A study with 80% power and 95% significance to detect a 35% reduction in the incidence of pneumonia compared to the placebo group will require 22079 child months per group37. Since each child will be followed for 18 months the study will require 1227 child per group. Assuming a 20% loss to follow up the study requires 1472 child per group. In order to facilitate randomization and allocation of staff we have rounded this figure to 1500 child per group.

Sample size for blood test as process measure:

50 children per group will give 80% power to detect a 50% reduction in the proportion of children with 1,25(OH)2D <8ng/ml (50% being conservative compared to the published literature29-32), assuming that this deficiency is about 60% in the placebo group (a conservative estimate).

ELIGIBILITY:
Inclusion Criteria:

1. 1 to 11 month old infants living in the study area
2. caretakers are willing to give consent to take part in the study

Exclusion Criteria:

1. the family is likely to migrate out of the study area within the next 18 months
2. the child has been diagnosed with rickets or known to have received a course of vitamin D treatment in the past 3 monDths.
3. Child with Kwashiorkor or Marasmus.

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3048 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
incidence of pneumonia | 18 months

SECONDARY OUTCOMES:
incidence of diarrhoea | 18 months
incidence of ricketts | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chandramohan, MBBS MSc PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Semira Manaseki-Holland, MRCP PhD, Principal Investigator — Agh Khan Health Services; Zulfiqar A Bhutta, MD, Principal Investigator — Aga khan University, Karachi; Zulf Mughal, MRCP, Principal Investigator — Manchester Childrens Hosptial
Locations (2):
- Afghanistan (2):
  - Aga Khan Health Services, Kabul, Kabul
  - Maywand Hospital, Kabul

REFERENCES:
- [Derived] Crowe FL, Mughal MZ, Maroof Z, Berry J, Kaleem M, Abburu S, Walraven G, Masher MI, Chandramohan D, Manaseki-Holland S. Vitamin D for Growth and Rickets in Stunted Children: A Randomized Trial. Pediatrics. 2021 Jan;147(1):e20200815. doi: 10.1542/peds.2020-0815. Epub 2020 Dec 18. PMID 33386335
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Aluisio AR, Maroof Z, Chandramohan D, Bruce J, Masher MI, Manaseki-Holland S, Ensink JH. Risk factors associated with recurrent diarrheal illnesses among children in Kabul, Afghanistan: a prospective cohort study. PLoS One. 2015 Feb 13;10(2):e0116342. doi: 10.1371/journal.pone.0116342. eCollection 2015. PMID 25679979
- [Derived] Manaseki-Holland S, Maroof Z, Bruce J, Mughal MZ, Masher MI, Bhutta ZA, Walraven G, Chandramohan D. Effect on the incidence of pneumonia of vitamin D supplementation by quarterly bolus dose to infants in Kabul: a randomised controlled superiority trial. Lancet. 2012 Apr 14;379(9824):1419-27. doi: 10.1016/S0140-6736(11)61650-4. Epub 2012 Apr 10. PMID 22494826